CLINICAL TRIAL: NCT07255248
Title: Hoffa's Fat Pad Impingement (HFPI): Saline Injection Verus Ultrasound Guided Cortisone Injection: A Randomized Trial in Adolescent Female Athletes
Brief Title: Hoffa's Fat Pad Impingement (HFPI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Julie Han, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00051842
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hoffa's Fat Pad Impingement
MeSH Terms: interventions — Methylprednisolone Acetate; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Saline Injection (Placebo Comparator): If you are randomized to the control group, you will receive a saline injection to the hoffa's fat pad at your visit. Saline injections are safe for the intended use of being a placebo injection. After your injection, you will be required to continue with physical therapy. You will be sent patient reported outcomes including quality of life, pain interference, symptoms and function, and level of activity at 4 weeks and 8 weeks following your injection.
  Interventions: Drug: Saline injection (Octreotide LAR placebo)
- Intervention Group: Corticosteroid Injection (Active Comparator): If you are randomized to the intervention group, you will receive an ultrasound guided corticosteroid injection to the hoffa's fat pad at your visit. Ultrasound guided corticosteroids injections are a common and approved procedure for this condition done at Boston Children's Hospital in the sports medicine clinic. You will be sent patient reported outcomes including quality of life, pain interference, symptoms and function, and level of activity at 4 weeks and 8 weeks following your injection.
  Interventions: Drug: methylprednisolone acetate and lidocaine

INTERVENTIONS:
Drug: methylprednisolone acetate and lidocaine — If you are randomized to the intervention group, you will receive an ultrasound guided corticosteroid injection to the hoffa's fat pad at your visit. Ultrasound guided corticosteroids injections are a common and approved procedure for this condition done at Boston Children's Hospital in the sports medicine clinic. You will be sent patient reported outcomes including quality of life, pain interference, symptoms and function, and level of activity at 4 weeks and 8 weeks following your injection.
  Arms: Intervention Group: Corticosteroid Injection
Drug: Saline injection (Octreotide LAR placebo) — If you are randomized to the control group, you will receive a saline injection to the hoffa's fat pad at your visit. Saline injections are safe for the intended use of being a placebo injection. After your injection, you will be required to continue with physical therapy. You will be sent patient reported outcomes including quality of life, pain interference, symptoms and function, and level of activity at 4 weeks and 8 weeks following your injection.
  Arms: Control Group: Saline Injection

SUMMARY:
The aim of the study is to investigate treatment outcomes for refractory anterior knee pain due to Hoffa's Fat Pad Impingement (HFPI) in young female athletes. Specifically, the study team will study pediatric female athletes with HFPI, and treatment outcomes of US-guided Hoffa's Fat Pad (HFP) corticosteroid injection compared to standard care (physical therapy, bracing, no injection) and saline injection. There will be two arms in this study, 1, a corticosteroid injection and physical therapy and 2, physical therapy and a saline injection. The intent of this study is to measure treatment outcomes, and the research team is not looking at the safety and effectiveness of the lidocaine-methylprednisolone mixture.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HFPI (defined as pain to palpation over the medial or lateral aspect of the infrapatellar fat pad, and/or positive hoffa test which is performed by exerting direct pressure over the infrapatellar fat pad as the knee is passively moved from flexion to extension; pain is positive hoffa test)
* Age 12-18 years
* Patients who identify as female
* Organized sports participation is defined as any adult-led game or sport in which three or more people play and/or practice together regularly in a league or association or an adult-led individual athletic activity. Non-organized sport is excluded such as free play.
* Xray and non-contrast MRI of the knee must have been completed for the symptomatic knee
* Must have completed physician-prescribed course of physical therapy for 6-8 weeks

Exclusion Criteria:

* History of patellar dislocation or subluxation, Ehlers-Danlos syndrome, patellar tendinitis/tendinosis, quadriceps tendinitis/tendinosis, medial plica syndrome, osteochondritis dessicans (OCD) of the knee, knee osteoarthritis, prior knee surgery
* Other concurrent knee derangement such as meniscus or ligament tears
* Radiographic evidence of bony abnormalities other than lateral patellar tilt, patella alta/baja, trochlear dysplasia
* MR positive for internal knee joint derangement, synovitis/inflammatory changes/effusion, OCD
* Patients receiving other knee injections during the study time period (i.e., viscosupplementation injection, Toradol injection)

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC Score) | From enrollment to 8 weeks after enrollment
  The IKDC is a patient-reported outcome measure on a 0-100 scale assessing knee function, symptoms, and sports activities, with higher scores indicating better function, and a lower score indicating low function.

SECONDARY OUTCOMES:
Peds Quality of Life Score (Peds-QL) | From enrollment to 8 weeks after enrollment
  The Pediatric Quality of Life Inventory (PedsQL) is a brief measure of health-related quality of life in children and young people. Scoring involves transforming a 0-4 Likert scale (0=never, 4=almost always) into a 0-100 scale by reverse scoring and linear transformation, where higher scores indicate better health-related quality of life and a lower score indicating low health-related quality of life (HRQL).
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form (PISF) | From enrollment to 8 weeks after enrollment
  The PISF is designed to measure the extent to which pain interferes with a person's: Work or household chores, Social activities, Enjoyment of life, and Physical activities. Each question has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. A higher score indicates higher pain levels and pain interference, and a lower score indicates lower pain interference.
Level of Activity per week | From enrollment to 8 weeks after enrollment
  Patients will report hours of activity per week during the study
Self-report pain flare post injection | 4 weeks post injection
  Patients will self-report any pain flares that occur 4 weeks after receiving the injection

CONTACTS AND LOCATIONS:
Overall Officials: Julie Han, M.D., Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
All IPD that will be shared will be de-identified and for manuscript and publishing purposes only. PHI data will not be accessible outside of the research team, and only de-identified data will be a part of the manuscript.
Time Frame: IPD will be analyzed for the manuscript, and all will be de-identified. This is approximately from the end of the study collection December 2027 to June 2028 for analysis.

REFERENCES:
- [Background] Katz NB, Tsitsilianos N, Nowak AS, Douglas SR, Tenforde AS, Borg-Stein J. Advanced Non-Operative Interventions for Anterior Knee Pain. Curr Rev Musculoskelet Med. 2024 Dec;17(12):589-615. doi: 10.1007/s12178-024-09930-x. Epub 2024 Nov 11. PMID 39527393
- [Background] House CV, Connell DA. Therapeutic ablation of the infrapatellar fat pad under ultrasound guidance: a pilot study. Clin Radiol. 2007 Dec;62(12):1198-201. doi: 10.1016/j.crad.2007.07.005. Epub 2007 Sep 14. PMID 17981168
- [Background] Bessette M, Saluan P. Patellofemoral Pain and Instability in Adolescent Athletes. Sports Med Arthrosc Rev. 2016 Dec;24(4):144-149. doi: 10.1097/JSA.0000000000000133. PMID 27811513
- [Background] Chung CB, Skaf A, Roger B, Campos J, Stump X, Resnick D. Patellar tendon-lateral femoral condyle friction syndrome: MR imaging in 42 patients. Skeletal Radiol. 2001 Dec;30(12):694-7. doi: 10.1007/s002560100409. Epub 2001 Sep 7. PMID 11810167
- [Background] Subhawong TK, Eng J, Carrino JA, Chhabra A. Superolateral Hoffa's fat pad edema: association with patellofemoral maltracking and impingement. AJR Am J Roentgenol. 2010 Dec;195(6):1367-73. doi: 10.2214/AJR.10.4668. PMID 21098197
- [Background] Feuerriegel GC, Marth AA, Frohlich S, Scherr J, Sporri J, Sutter R. Superolateral Hoffa fat pad edema in adolescent competitive alpine skiers: temporal evolution over 4 years and risk factors. Insights Imaging. 2024 Feb 16;15(1):52. doi: 10.1186/s13244-024-01633-8. PMID 38365902
- [Background] Mills MK, Allen H. Knee Plical Pathology and Impingement Syndromes. Magn Reson Imaging Clin N Am. 2022 May;30(2):293-305. doi: 10.1016/j.mric.2021.11.008. Epub 2022 Apr 13. PMID 35512891
- [Background] Eymard F, Chevalier X. Inflammation of the infrapatellar fat pad. Joint Bone Spine. 2016 Jul;83(4):389-93. doi: 10.1016/j.jbspin.2016.02.016. Epub 2016 Apr 7. PMID 27068617
- [Background] Dragoo JL, Johnson C, McConnell J. Evaluation and treatment of disorders of the infrapatellar fat pad. Sports Med. 2012 Jan 1;42(1):51-67. doi: 10.2165/11595680-000000000-00000. PMID 22149697
- [Background] Abelleyra Lastoria DA, Benny CK, Hing CB. Predisposing factors for Hoffa's fat pad syndrome: a systematic review. Knee Surg Relat Res. 2023 Jun 9;35(1):17. doi: 10.1186/s43019-023-00192-4. PMID 37296488